CLINICAL TRIAL: NCT04369378
Title: Effectiveness of Using a Meditation App in Reducing Anxiety and Improving Well-being During the Covid-19 Pandemic
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lake Erie College of Osteopathic Medicine (Other)
Responsible Party: Principal Investigator, Diana Speelman, Director of Research, Associate Professor of Biochemistry, Lake Erie College of Osteopathic Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 27-126
Record Dates: First submitted 2020-04-24; First posted 2020-04-30 (Actual); Last update posted 2021-08-30 (Actual); Status verified 2021-08

CONDITIONS: Anxiety; Well-being
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial: adults randomly assigned to daily use of a meditation app for 30 days or control group (no usage of meditation app).
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Meditation app group (Experimental): Participants will also be given access to the mindfulness app (Insight Timer), and instructed to use it for 10 min daily for 30 days. Two days before the end of the 30 day intervention period, participants will be sent a link to a Google Form for the post-intervention survey and will be asked to complete the survey within the next 3 days. Two months after the conclusion of the 30 day intervention period (90 days after study began), participants will be sent a link to a Google Form for another post-intervention survey, and asked to complete it within 5 days.
  Interventions: Behavioral: Meditation app usage
- Control group (No Intervention): Participants will be in the no intervention period for 30 days. Two days before the end of the 30 day no intervention period, participants will be sent a link to a Google Form for the post-intervention survey and will be asked to complete the survey within the next 3 days. After this 30 day no intervention period, participants are invited to use the Insight Timer app if they so choose. Two months after the conclusion of the 30 day no intervention period (90 days after study began), participants will be sent a link to a Google Form for another post-intervention survey, and asked to complete it within 5 days.

INTERVENTIONS:
Behavioral: Meditation app usage — Investigators will confirm eligibility of applicants, enroll participants in the study and provide an identification number for de-identification of the data, and provide a list of mental health resources to participants. Participants will then be sent a link to a Google Form for the pre-intervention survey, to be completed prior to first use of the mindfulness app. Participants will also be given access to the mindfulness app (Insight Timer), and instructed to use it for 10 min daily for 30 days. Two days before the end of the 30 day intervention period, participants will be sent a link to a Google Form for the post-intervention survey and will be asked to complete the survey within the next 3 days. Two months after the conclusion of the 30 day intervention period, participants will be sent a link to a Google Form for another post-intervention survey, and asked to complete it within 5 days.
  Arms: Meditation app group

SUMMARY:
This interventional study will investigate the effect of daily use of a mindfulness app on measures of participant anxiety, well-being, and future outlook during the Covid-19 pandemic, by comparing pre-intervention survey responses to post-intervention survey responses.

DETAILED DESCRIPTION:
Question 1: Can 30 days of daily use of a mindfulness app during the Covid-19 pandemic reduce anxiety and improve general well-being and future outlook? Outcomes measured: Pre- and post-intervention surveys to assess well-being and anxiety (primary outcomes), future outlook, hopefulness, and sleep habits (secondary outcomes). Many of these survey questions come from well-validated surveys (WHO-5 Well-being survey, GAD7 Anxiety survey). Post intervention surveys will be administered at the end of the 30d intervention, as well as 2 months after the completion of the 30d intervention.

Question 2: Can 30 days of daily use of a mindfulness app during the Covid-19 pandemic improve nutritional habits? Outcomes measured: Pre- and post-intervention surveys to assess general nutrition habits, including frequency of consuming whole foods (fruits, vegetables, whole grains) and frequency of consuming prepared meals (secondary outcomes). Post intervention surveys will be administered at the end of the 30d intervention, as well as 2 months after the completion of the 30d intervention.

Question 3: Will study participants be more likely to continue to use the mindfulness app after completion of the study? Outcomes measured: Post-intervention survey administered at the end of the 30d intervention will be used to assess likelihood to continue using app and frequency of anticipated continued use. The post-intervention survey administered 2 months after the completion of the 30d intervention will ask if participants continued to use the app, and the frequency of use (secondary outcomes).

ELIGIBILITY:
Inclusion Criteria:

* Participants must be 18 or older. Inclusion criteria are access to a smartphone and ability to download the mindfulness app, fluency in English, and the ability to complete surveys independently.

Exclusion Criteria:

* Exclusion criteria include current regular use of a mindfulness or meditation app, regular practice of mindfulness or meditation, regular therapy sessions, inability to complete surveys independently, or any mental health restrictions that would prevent them from participating.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2020-08-19 (Actual); Primary Completion 2021-04-28 (Actual); Study Completion 2021-08-26 (Actual)

PRIMARY OUTCOMES:
Anxiety | Immediate post-intervention (compare with pre-intervention data)
  Assessed by survey questions (in part adapted from GAD7)
Well-being | Immediate post-intervention (compare with pre-intervention data)
  Assessed by survey questions (in part adapted from WHO-5)

SECONDARY OUTCOMES:
Future outlook & hopefulness | Immediate post-intervention (compare with pre-intervention data)
  Assessed by survey questions
Sleep habits | Immediate post-intervention (compare with pre-intervention data)
  Assessed by survey questions
Nutrition habits | Immediate post-intervention (compare with pre-intervention data)
  Assessed by survey questions (frequency of consuming whole foods and prepared meals)
Meditation app continued usage | Immediate post-intervention (compare with pre-intervention data)
  Assessed by survey questions (anticipated and actual continued usage of app)
Anxiety | 2 months post-intervention (compare with pre-intervention, immediate post-intervention data)
  Assessed by survey questions (in part adapted from GAD7)
Well-being | 2 months post-intervention (compare with pre-intervention, immediate post-intervention data)
  Assessed by survey questions (in part adapted from WHO-5)
Future outlook & hopefulness | 2 months post-intervention (compare with pre-intervention, immediate post-intervention data)
  Assessed by survey questions
Sleep habits | 2 months post-intervention (compare with pre-intervention, immediate post-intervention data)
  Assessed by survey questions
Nutrition habits | 2 months post-intervention (compare with pre-intervention, immediate post-intervention data)
  Assessed by survey questions (frequency of consuming whole foods and prepared meals)
Meditation app continued usage | 2 months post-intervention (compare with immediate post-intervention data)
  Assessed by survey questions (anticipated and actual continued usage of app)

CONTACTS AND LOCATIONS:
Overall Officials: Diana Speelman, PhD, Principal Investigator — Lake Erie College of Osteopathic Medicine
Locations (1):
- LECOM, Erie, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified participant data will be reported as individual data points, as well as means +/- SD or medians with quartiles.
Supporting Information: Study Protocol, SAP
Time Frame: Upon publication of findings
Access Criteria: Upon written request to corresponding author on publication

REFERENCES:
- [Derived] O'Donnell KT, Dunbar M, Speelman DL. Effectiveness of using a meditation app in reducing anxiety and improving well-being during the COVID-19 pandemic: A structured summary of a study protocol for a randomized controlled trial. Trials. 2020 Dec 9;21(1):1006. doi: 10.1186/s13063-020-04935-6. PMID 33298117